CLINICAL TRIAL: NCT00337558
Title: Solifenacin Succinate in a Flexible Dose Regimen With Simplified Bladder Training Versus Solifenacin Succinate in a Flexible Dose Regimen Alone in a Prospective, Randomized, Parallel Group, Overactive Bladder Symptom Study
Brief Title: A Study of Solifenacin With Bladder Training Versus Solifenacin Alone in Patients With Overactive Bladder (SOLAR)
Acronym: SOLAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 905-EC-003
Record Dates: First submitted 2006-06-14; First posted 2006-06-16 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Overactive Bladder; Urinary Incontinence; Urge Incontinence
Keywords: treatment outcomes; Overactive bladder; Solifenacin succinate; urinary incontinence; urge incontinence; frequency
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence; Urinary Incontinence, Urge | interventions — Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Solifenacin succinate
  Interventions: Drug: Solifenacin succinate
- 2 (Experimental): Solifenacin succinate and simplified bladder training
  Interventions: Behavioral: Simplified bladder training

INTERVENTIONS:
Drug: Solifenacin succinate — tablet
  Other Names: YM905
  Arms: 1
Behavioral: Simplified bladder training — Instructions
  Arms: 2

SUMMARY:
This study will look at a drug for OAB (solifenacin) in combination with a non drug treatment (bladder training) compared to the drug on its own. The study will compare the symptoms of OAB by assessing patient diaries and other patient reported outcomes.

DETAILED DESCRIPTION:
Subjects are screened between day -14 and day -1.

At day 0 subjects will enter a randomized, parallel group study. After fulfilling all selection criteria, subjects will be randomized to one of two treatment arms, solifenacin 5mg with bladder training or solifenacin 5mg alone. After 8 weeks of treatment subjects will be sub divided; subjects on solifenacin 5mg with bladder training will be given the option to increase dose and be divided into solifenacin 5mg with bladder training or solifenacin 10mg with bladder training. Subjects on solifenacin alone, will also be given the option to increase dose and be divided into solifenacin 5mg alone and solifenacin 10mg alone.

There are 5 visits in total: visit 1(screening), visit 2 (randomisation), visit 3 (week 4), visit 4 (week 8), telephone visit (week 12) and visit 5 (week 16)

All subjects receive medication in the form of solifenacin succinate 5mg tablets (two tablets for 10mg) (Company code: YM905, Company serial number: RVG29151)

Subjects randomized to bladder training will receive a single sheet of instructions for bladder training.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of overactive bladder (including urinary frequency, urgency with/without urge incontinence) for> 3 months

Exclusion Criteria:

* Clinically significant outflow obstruction
* Significant post void residual volume
* Significant stress incontinence or mixed stress/urge incontinence where stress is the predominant factor as determined by the investigator.
* Patient with a neurological cause for abnormal detrusor activity.
* Evidence of a symptomatic urinary tract infection, chronic inflammation such as interstitial cystitis, bladder stones, previous pelvic radiation therapy or previous or current malignant disease of the pelvic organs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 643 (Actual)
Dates: Start 2006-05; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean number of micturitions per 24 hours after 8 weeks | 8 weeks

SECONDARY OUTCOMES:
Change from baseline in mean number of micturitions per 24 hours after 16 weeks | 16 weeks
Change from baseline in mean urgency frequency per 24 hours | 8 and 16 weeks
Change from baseline in mean number of incontinence and urge incontinence episodes per 24 hours | 8 and 16 weeks
Change from baseline in number of pads used | 8 and 16 weeks
Incidence and severity of adverse events | 8 and 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Astellas Medical Affairs Europe, Principal Investigator — University Hospital, Lund, Sweden
Locations (56):
- Australia (6):
  - Kogarah, New South Wales
  - Randwick, New South Wales
  - Auchenflower, Queensland
  - Clayton, Victoria
  - Concord
  - Parkville
- Belgium (6):
  - Antwerp
  - Brussels
  - Ghent
  - Kortrijk
  - La Louvière
  - Sint-Truiden
- Czechia (5):
  - Jihlava
  - Liberec
  - Olomouc
  - Pilsen
  - Prague
- France (12):
  - Annecy
  - Arras
  - Bordeaux
  - Landerneau
  - Marseille
  - Paris
  - Rouen
  - Saint-Louis
  - Thionville
  - Toulouse
  - Valenciennes
  - Vernon
- Hungary (4):
  - Budapest
  - Kecskemét
  - Nyíregyháza
  - Tatabánya
- Italy (6):
  - Bari
  - Cinisello Balsamo
  - Como
  - Genova
  - Milan
  - Naples
- Netherlands (4):
  - Leiden
  - Roermond
  - Tilburg
  - Zwijndrecht
- Warsaw, Poland
- Russia (2):
  - Moscow
  - Saint Petersburg
- Spain (8):
  - Avilés
  - Burgos
  - Madrid
  - Manacor
  - Marbella
  - Santander
  - Santiago de Compostela
  - Seville
- Turkey (Türkiye) (2):
  - Ankara
  - Istanbul

REFERENCES:
- [Background] Mattiasson A, Masala A, Morton R, Bolodeoku J; SOLAR Study Group. Efficacy of simplified bladder training in patients with overactive bladder receiving a solifenacin flexible-dose regimen: results from a randomized study. BJU Int. 2010 Apr;105(8):1126-35. doi: 10.1111/j.1464-410X.2009.08910.x. Epub 2009 Oct 10. PMID 19818077
- [Derived] Funada S, Yoshioka T, Luo Y, Sato A, Akamatsu S, Watanabe N. Bladder training for treating overactive bladder in adults. Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD013571. doi: 10.1002/14651858.CD013571.pub2. PMID 37811598